CLINICAL TRIAL: NCT06622161
Title: Automated Oxygen Control in Preterm Babies on Respiratory Support: A Randomized Cross Over Study
Brief Title: Automated Versus Manual Oxygen Control in Preterm Babies on Respiratory Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Ali Shabbir Hussain, Assistant Professor & Section Head NICU, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10189
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Preterm
Keywords: Respiratory; Hypoxia; Hyperoxia; Oxygen saturation; Target range
MeSH Terms: conditions — Premature Birth; Hypoxia; Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- "automated oxygen," (Other): Preterm babies will be kept on the SLE 6000 ventilator for 12 hours, where an automated oxygen device called "oxygenie" will be used to automatically adjust FiO2 to keep SpO2 within the target range. After 12 hours, the other group will be kept on this arm for 12 hours.
  Interventions: Device: automated oxygen vs manual oxygen
- "manual oxygen" (Other): Preterm babies will be kept on the SLE 6000 ventilator for 12 hours, where manual FiO2 adjustment by the bedside staff nurse will be used to keep SpO2 within the target range. After 12 hours, the other group will be kept on this arm for 12 hours.
  Interventions: Device: automated oxygen vs manual oxygen

INTERVENTIONS:
Device: automated oxygen vs manual oxygen — Patient characteristics, ventilator, and blood gas parameters at the time of study will be shown in Tabular form. At the start of the study, half of the babies will be randomly assigned to a manual 12-hour period where a bedside nurse will adjust the FiO2 of the baby according to SpO2 levels, and half of the babies to an automated 12-hour period where Oxygenie will adjust FiO2 according to target SpO2 levels. After 12 hours, they will be shifted to contralateral intervention. The ventilator parameters (peak inspiratory pressure, positive end expiratory pressure, and rate) will be compared between the automated and manual 12-hour periods. The amount of time spent within different ranges of SpO2 will also be measured and shown in tabular form.

SUMMARY:
Babies admitted in the NICU (neonatal intensive care unit) frequently need supplemental oxygen to keep their oxygen saturation (SpO2) in target range (TR). Hypoxia and hyperoxia episodes should be avoided while working toward this goal. Preterm babies are particularly vulnerable to abnormal oxygen levels, and adverse effects of hyperoxia and oxygen toxicity may result in retinopathy of prematurity and bronchopulmonary dysplasia. Similarly, mortality may rise due to hypoxic events. In routine practice, the SpO2 target is usually achieved by manual adjustment of FiO2 (fraction of inspired oxygen), but it usually does not accomplish the desired SpO2 target, leading to episodes of hyperoxia and hypoxia and increased risk of complications. A study was conducted in multiple centers involving extremely preterm babies, the results of which depicted that the babies on manual control of FiO2 spent only 48% of their time with SpO2 in the target range, 16% below the target range, and 36% above it. The compliance of the SpO2 target range was also variable in these centers. There is a need to improve compliance by using automated oxygen control systems.

At the Aga Khan University Hospital (AKUH) investigators have included SLE 6000 (SLE, Croydon, UK) ventilators in their NICU (neonatal intensive care unit) which have automated oxygen control device "Oxygenie" that continuously adjusts FiO2 (fraction of inspired oxygen) of the patient to keep SpO2 in the target range, avoiding abnormal oxygen levels. This also reduces the workload on staff and improves patient care. Investigators usually put preterm babies on these ventilators so that SpO2 can be kept most of the time in the target range. When the OxyGenie and SpO2 monitoring are added to the SLE 6000 ventilator, it becomes possible to accurately regulate and deliver closed loop oxygen to preterm infants. This automated oxygen control system limits episodes of both hypoxia and hyperoxia by using the VDL 1.1 algorithm that uses an adaptive Proportional-Integral-Derivative (PID) algorithm to control the FiO2 adjustments in response to changes in SpO2. This keeps SpO2 within a target range (TR) which user selects. A randomized crossover trial comparing two devices for automated oxygen control in preterm infants included the SLE 6000 ventilator as one of its devices.

DETAILED DESCRIPTION:
Investigators will conduct a radomized cross-over trial. 24 Preterm babies will be sampled, and to account for attrition, 26 preterm babies will be enrolled. Preterm babies born at less than 37 weeks of gestation will be included in the study. For each of the twelve-hour periods, they will be randomized to either manually controlled oxygen or automated oxygen control. After 12-hour periods, they will be shifted to alternate interventions. The total duration will be 24 hours. Written consent will be obtained from the parent/guardian before recruitment.

Block randomization will be done to randomize the babies. SLE 6000 ventilators will be used, and settings will be adjusted by the clinical team as per the clinical condition of the baby.

The Radical neonatal pulse oximeter (Masimo) is used to automatically adjust FiO2 in order to maintain SpO2 within a designated target range. Before turning on oxygen, FiO2 is manually adjusted to achieve SpO2 in the target range. Once stable SpO2 is achieved in TR, oxygen is turned on, which then adjusts FiO2 to keep SpO2 within target range. The FiO2 changes and their frequency are determined by the SpO2 trend, whether the SpO2 is above, below, or within the target range, and all changes are proportionate to the baseline FiO2 level. The pulse oximeter's settings will include normal sensitivity, an average time of 2-4 seconds, a 20-second alarm delay, and an alarm limit of 89% and 95% SpO2. Whenever feasible, the right wrist is used to apply the Masimo neonatal probe. The user will be advised on screen if the SpO2 signal will be lost. Oxygenie would display in blue, waiting for a signal, and would remain on the current FiO2 value for the first 60 seconds. After this point, if the SpO2 is within TR, it will continue at the current FiO2 level. If the SpO2 is above the TR and the FiO2 is 10% above the reference range, it will slowly decrease to the reference value. If SpO2 is below TR and FiO2 is more than 5% below the reference FiO2, then it will slowly increase to the reference level. The reference FiO2 value is updated every 30 minutes and is based on the last 60-minute average.

ELIGIBILITY:
Inclusion Criteria:

Investigators will include premature babies (born before 37 weeks of pregnancy) who are on SLE 6000 ventilator, and require additional oxygen therapy or respiratory support due to respiratory dysfunction.

Preterm babies will be included in the study if they will meet all the following criteria:

* Receiving respiratory support via mechanical ventilation, either non-invasive or invasive
* Receiving supplemental oxygen at the time of inclusion
* Written informed parental consent

Exclusion Criteria:

* Major Congenital Anomalies such as neural tube defects, neuromuscular disorders, congenital heart diseases, syndromic babies, and so forth.
* Resuscitation and termination of mechanical ventilation during the study
* Withdrawal of parent consent

Max Age: 13 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Percentage of time with SpO2 within the target range | 12 hours on each arm
  The primary outcome measure of time with SpO2 within the target range of 90-94% will be compared between automated and manual period.

SECONDARY OUTCOMES:
Percentage of time with SpO2 above the target range and below the target range | 12 hours on each arm
  The percentage of time with SpO2 above the target range (>94% and ≥98%) with FiO2 of >0.21 and below the target range (<90% and <80%) will be compared between both interventions.
SpO2 fluctuations below 80% and 98% or above, and episodes of prolong hypoxia and hyperoxia | 12 hours on each arm
  Between automated and routine care, we'll also track the number and median duration of SpO2 fluctuations below 80% and 98% or above, as well as episodes of prolong hypoxia and hyperoxia of one and three minutes
Median FiO2 values and median number of manual adjustments of FiO2 | 12 hours on each arm
  Median FiO2 values and median number of manual adjustments of FiO2 will be compared between both automated and manual control periods
% of Time with SpO2 in Target range (90-94%), <90%, and > 94%, with and without use of sedative and respiratory stimulant medications | 12 hours on each arm
  The percentage of time with SpO2 in the target range (90-94%), below (<90%), and above (>94%) the target range when FiO2 > 21%, in babies with and without sedative and respiratory stimulant medication use (e.g., Morphine, Caffeine, etc.) will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shabbir Hussain, Principal Investigator — Aga Khan University Hospital, Karachi, Pakistan
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston ED, Boyle B, Juszczak E, King A, Brocklehurst P, Stenson BJ. Oxygen targeting in preterm infants using the Masimo SET Radical pulse oximeter. Arch Dis Child Fetal Neonatal Ed. 2011 Nov;96(6):F429-33. doi: 10.1136/adc.2010.206011. Epub 2011 Mar 6. PMID 21378398
- [Background] van Kaam AH, Hummler HD, Wilinska M, Swietlinski J, Lal MK, te Pas AB, Lista G, Gupta S, Fajardo CA, Onland W, Waitz M, Warakomska M, Cavigioli F, Bancalari E, Claure N, Bachman TE. Automated versus Manual Oxygen Control with Different Saturation Targets and Modes of Respiratory Support in Preterm Infants. J Pediatr. 2015 Sep;167(3):545-50.e1-2. doi: 10.1016/j.jpeds.2015.06.012. Epub 2015 Jul 2. PMID 26144575
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Background] Stenson B, Brocklehurst P, Tarnow-Mordi W; U.K. BOOST II trial; Australian BOOST II trial; New Zealand BOOST II trial. Increased 36-week survival with high oxygen saturation target in extremely preterm infants. N Engl J Med. 2011 Apr 28;364(17):1680-2. doi: 10.1056/NEJMc1101319. No abstract available. PMID 21524227
- [Background] Laptook AR, Salhab W, Allen J, Saha S, Walsh M. Pulse oximetry in very low birth weight infants: can oxygen saturation be maintained in the desired range? J Perinatol. 2006 Jun;26(6):337-41. doi: 10.1038/sj.jp.7211500. PMID 16598294
- [Background] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549
- [Background] Salverda HH, Oldenburger NJ, Rijken M, Pauws SC, Dargaville PA, Te Pas AB. The effect of automated oxygen control on clinical outcomes in preterm infants: a pre- and post-implementation cohort study. Eur J Pediatr. 2021 Jul;180(7):2107-2113. doi: 10.1007/s00431-021-03982-8. Epub 2021 Feb 23. PMID 33619593
- [Background] Dargaville PA, Sadeghi Fathabadi O, Plottier GK, Lim K, Wheeler KI, Jayakar R, Gale TJ. Development and preclinical testing of an adaptive algorithm for automated control of inspired oxygen in the preterm infant. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F31-F36. doi: 10.1136/archdischild-2016-310650. Epub 2016 Sep 15. PMID 27634820
- [Background] Gajdos M, Waitz M, Mendler MR, Braun W, Hummler H. Effects of a new device for automated closed loop control of inspired oxygen concentration on fluctuations of arterial and different regional organ tissue oxygen saturations in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F360-F365. doi: 10.1136/archdischild-2018-314769. Epub 2018 Aug 28. PMID 30154236
- [Background] Salverda HH, Cramer SJE, Witlox RSGM, Gale TJ, Dargaville PA, Pauws SC, Te Pas AB. Comparison of two devices for automated oxygen control in preterm infants: a randomised crossover trial. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):20-25. doi: 10.1136/archdischild-2020-321387. Epub 2021 Jun 10. PMID 34112721
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Reynolds PR, Miller TL, Volakis LI, Holland N, Dungan GC, Roehr CC, Ives K. Randomised cross-over study of automated oxygen control for preterm infants receiving nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F366-F371. doi: 10.1136/archdischild-2018-315342. Epub 2018 Nov 21. PMID 30464005
- [Background] Salverda HH, Cramer SJE, Witlox RSGM, Dargaville PA, Te Pas AB. Automated oxygen control in preterm infants, how does it work and what to expect: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2021 Mar;106(2):215-221. doi: 10.1136/archdischild-2020-318918. Epub 2020 Jul 30. PMID 32732378
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Derived] Aamir Yousuf HM, Hussain AS, Schmolzer GM, Hoodbhoy Z, Munir R, Rizvi A, Khan U. Automated oxygen control in preterm babies on respiratory support: protocol for a randomised crossover trial. BMJ Paediatr Open. 2025 May 14;9(1):e003210. doi: 10.1136/bmjpo-2024-003210. PMID 40374283
- See also: Automated Oxygen Delivery in Neonatal Intensive Care — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9257066/